CLINICAL TRIAL: NCT05983341
Title: Relapse of VAD Infections After Discontinuation of Anti-infective Therapies in Children.
Brief Title: Complications in Pediatric Mechanical Circulatory Assistance: Evaluation of Infection Management.
Acronym: VADINFECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0790
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Implant Infection
Keywords: Berlin Heart EXCOR; pediatric; VAD infections; Heart Failure; implanted material infection.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children (<18 years old) with Berlin Heart EXCOR assisting device.

SUMMARY:
End-stage heart failure in children is a rare cause of infant mortality. The most frequent cause is dilated cardiomyopathy, often of undetermined origin, which can lead to cardiogenic shock refractory to standard medical treatment. In such cases, it is essential to resort to exceptional means, available at tertiary care hospitals such as in Lyon. The therapeutic means includes long-term circulatory assistance (VAD). This type of circulatory assistance is becoming increasingly used in view of the shortage of heart transplants. Indeed, the average waiting time on the paediatric transplant list varies from 3 months to over a year for children under 5. Berlin Heart EXCOR (BHE) is the only long-term support available for children (2). It is a pulsatile para-corporeal assisting device with percutaneous cannulas.

Despite technical and medical advances in circulatory support, the presence of foreign material is frequently complicated by infection. Infection is a major cause of morbidity and mortality in this population. It is most often of nosocomial origin, linked to central line infections. The germs associated with these infections are mainly bacteria, with a small proportion of fungi. The most common pathogens are multi-resistant gram-positive bacteria, which colonize the skin, adhere to the implanted equipment and create biofilms. Infections have a major impact on the morbidity and mortality of patients undergoing mechanical assistance, with an increased risk of thrombo-embolic events and difficulty in managing anticoagulation, secondary to inflammation.

DETAILED DESCRIPTION:
There are few literatures on the management of infections under mechanical assistance. Current ISHLT (International Society for Heart and Lung Transplantation) recommendations are based on expert opinion and observational studies. Actual recommendations are long-term anti-infective therapy, even up to the time of transplantation in the case of assistance-specific or assistance-associated infections.

At the Hospices Civils de Lyon, BH-assisted patients awaiting transplantation are cared for in the paediatric cardiac intensive care unit (PCICU). Infections are managed jointly with the infectious diseases team, through weekly consultations and RCP. The management strategy is directed towards the rational use of antibiotics and antifungals, to limit the impact of broad-spectrum, long-term antibiotic therapy on the microbiological environment and on the patient. The duration of anti-infective therapy is limited on the basis of clinical and biological criteria. In some cases, recurrence of the infectious episode may occur.

This study will provide information on the therapeutic strategy for VAD infections.

ELIGIBILITY:
* Inclusion Criteria * :

  * Age < 18years old
  * Berlin Heart EXCOR implantation
* Exclusion Criteria * :

  * None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Heart failure pediatric patients in need of ventricular assisting device
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Relapse of infection defined as an infection with an identical from a previous infectious episode germ (microbiological characterization and similar resistance profile). | From time of Berlin Heart EXCOR implantation to up to 6 months after heart transplantation.
  Clinical and microbiological diagnosis of a relapse of infection with the same germ after discontinuation of anti-infective therapy in the context of a specific or assistance-related infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mere eEnfant, Bron, Auvergne-Rhône-Alpes, France